CLINICAL TRIAL: NCT03430804
Title: Transvaginal Sonographic Measurement of Cervical Length Versus Bishop Score in Induction of Labour at Term for Prediction of Caesarean Delivery
Brief Title: Transvaginal Sonographic Measurement of Cervical Length Versus Bishop Score in Induction of Labour for Prediction of Caesarean Delivery.
Status: Completed | Type: Observational
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Mohamed Adel Mazroa, Dr resident of obstetrics and gynecology, Ain Shams University
Other Study IDs: Asu-August 2017
Record Dates: First submitted 2018-01-31; First posted 2018-02-13 (Actual); Last update posted 2018-02-14 (Actual); Status verified 2018-02

CONDITIONS: Failed Induction; Cervical Dystocia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Single gruop320 parturients: Measurement of cervical length and digital examination of Bishop score in 320 women undergoing induction of labour will be carried out in ain shams university maternity hospital.
  Interventions: Other: Bishop score calculation of modified Bishop score in numbers by digital vaginal examination

INTERVENTIONS:
Other: Bishop score calculation of modified Bishop score in numbers by digital vaginal examination — Measurement of cervical length by transvaginal ultrasound and digital examination of Bishop score in 320 parturients undergoing labour induction at term
  Other Names: cervical length measuring cervical length by trans-vaginal ultrasound

SUMMARY:
Transvaginal sonographic measurement of cervical length versus Bishop score in labour induction at term for prediction of Caesarean delivery. This study is prospective study. This study will be carried out in Ain-shams maternity hospital. Sample size of 320 parturients.

DETAILED DESCRIPTION:
Patients and Methods

Study design:

This study is prospective study, comparative clinical trial for a test against a gold standard with blinding of the evaluator

Study setting:

This study will be carried out in Ain-Shams university maternity hospital.

Methods:

* All patients recruited were given an oral consent.
* All patients were subjected to the following:

History of the patient:

* Detailed and careful history was taken from the patient as the following:

  1. Personal history: name, age, occupation, residence and special habit of medical importance.
  2. Obstetric history: including last menstrual period, Gestation age and regular Antenatal care.
  3. Past history: including any medical disorder e.g. Diabetes mellitus, hypertension or any surgical procedure
  4. History of present pregnancy: duration of pregnancy from last menstrual period, any complications occurred or any medication used during pregnancy.

     Examination of the patient:

  <!-- -->

  1. General examination: as regard level of consciousness, vital data, and complexion.
  2. Abdominal examination: as regard fundal level, lie of the fetus, detection of any uterine contractions and fetal heart rate.
  3. Pelvic Examination: as regard pelvic capacity, presenting part, presence of rupture of membranes and cervical assessment as regard cervical dilation, station and presenting part.
* Investigations. Complete blood count , Rh, transvaginal ultra sound and non-stress test.
* All patients had vaginal examination for assessing the (Bishop Score,1964) before induction of labour.
* All women had transvaginal ultrasound for assessment of cervical length using (median digital GAIA) Ultrasonic machine.

Protocol of transvaginal ultrasound will be done as follow:

1. Patient will be asked to void.
2. Vaginal probe will be inserted using direct visualization with K-Y gel.
3. Identification of bladder, amniotic fluid and fetal presenting part.
4. Identification of abnormal findings as placenta pervia or absence of fetal heart motion.
5. Identification of midline sagittal plane of the cervix and looking in the proximal one third of the image for the internal os then pulling back the probe until the lightest touch provides good image of the cervical canal and moving the probe slightly to get the best long axis of the cervix then measuring the cervical length by placing the calipers appropriately and recording the distance between internal and external cervical os.

   * Transvaginal ultrasound will be done to assess cervical length using medison sonoace 8800 (median digital GAIA) ultrasound machine equipped with a 7.5 m hertz by vaginal probe in Ain-Shams University Maternity Hospital.
   * Induction of labour will be done using intravaginal misoprostol (25 microgram) then digital examination will be made 6 h after the first intravaginal administration; if necessary, 3 doses were given at 6 hours interval. External Cardiotocography will be regularly performed to monitor the condition of the fetus.
   * Continuous Cardiotocography will be used in all cases. If necessary, amniotomy will be performed. Intravenous oxytocin administration will be started when there is an arrest of dilatation, starting at 1milli-international unit/minute and increasing 1 mIU every 30 min as necessary. For analgesia, intramuscular pethidine will be offered.
   * Caesarean delivery will be done due to pathological fetal heart rate trace, arrest the fetal head for at least one hour despite adequate uterine contractions.

ELIGIBILITY:
Inclusion Criteria:

* 1. Age (18-35) years. 2. Singleton pregnancy. 3. (37-42) weeks gestation. 4. Living fetus. 5. Cephalic presentation. 6. Absence of active labour. 7. No contraindication to vaginal delivery. 8. Average amount of clear liquor. 9. No history of uterine scar (myomectomy or previous C.S(.

Exclusion Criteria:

* 1. Malpresentation. 2. Major fetal congenital anomalies as hydrocephalous & dead fetus. 3. Patient received any pre induction ripping methods for example: (Acetic Acid-Prostaglandins).

  4. Any medical history contraindicating vaginal delivery. 5. Assessment meconium staining to liquor or any evidence of chorioamnionitis. 6. Previous uterine surgery. 7. Multiple gestations. 8. Women with allergy to prostaglandins.

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Single group 320 parturients udergoing induction of labour at term
Sampling Method: Probability Sample
Enrollment: 320 (Actual)
Dates: Start 2017-08-14 (Actual); Primary Completion 2017-12-14 (Actual); Study Completion 2018-01-12 (Actual)

PRIMARY OUTCOMES:
Cervical length | 24 hours
  median cervical length measured by transvaginal ultrasound in centimetres.
Bishop score | 72
  median Bishop score assessed by digital vaginal examination as follows: Cervical dilatation in centimeters will be given a score of zero if closed, a score of 1 if 1-2 cm dilated, a score of 2 if 3-4 cm dilated and a score of 3 if 5 cm or more dilatation.
  Effacement of the cervix will be given a score of zero if 0-30%, a score of 1 if 40-50%, a score of 2 if 60-70% and a score of 3 if 80% or more.
  Station of fetal head will be given a score of zero if -3, a score of 1 if -2, a score of 2 if -1 to zero and a score of 3 if 1 or more.
  Consistency of the cervix will be given a score of zero if firm, a score of 1 if medium and a score of 2 if soft.
  Position of the cervix will be given a score of zero if posterior, a score of 1 if mid position and a score of 2 if anterior. So, a total score (sum of all scores) of zero at a minimum to 10 at a maximum can be estimated.
  Note that a score more than 10 means patient is in labor not needing induction of labor.

CONTACTS AND LOCATIONS:
Locations (1):
- Mohamed adel mazroa, Tanta, Egypt